CLINICAL TRIAL: NCT06217185
Title: The Efficacy and Safety of Pyrotinib, Trastuzumab Combined With Taxanes in the Treatment of Early Trastuzumab-treated HER2+ Advanced Breast Cancer (ABC).
Brief Title: The Efficacy and Safety of Pyrotinib, Trastuzumab Combined With Taxanes in the Treatment of Trastuzumab-treated HER2+ Advanced Breast Cancer (ABC).
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-101
Record Dates: First submitted 2023-12-24; First posted 2024-01-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: HER2-positive Breast Cancer; Advanced Breast Cancer
MeSH Terms: interventions — pyrotinib; Trastuzumab; Taxoids; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Pyrotinib, Trastuzumab Combined With Taxanes
  *When taxane drugs are discontinued (after completing 6-8 cycles of treatment or due to intolerance), the therapy can be continued with the combination of metronomic capecitabine and trastuzumab, along with pyrotinib.
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Taxanes; Drug: Capecitabine

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400mg qd po continuously
Drug: Trastuzumab — For Trastuzumab, the loading dose for the first treatment cycle is 8 mg/kg, and for subsequent cycles, 6 mg/kg. It is to be used once every three weeks
Drug: Taxanes — Taxanes: Usual clinical dose is administered, in a 21-day cycle.
Drug: Capecitabine — Capecitabine: 650mg/m2 each time, given twice daily

SUMMARY:
This is a multi-center real-world study, in which patients who meet the inclusion criteria will receive treatment with Pyrotinib + Trastuzumab + Taxanes. Taxanes will be used for 6-8 cycles or discontinued due to intolerable Adverse Events (AEs), after which Capecitabine will be used for rhythmic chemotherapy combined with Pyrotinib + Trastuzumab. The aim is to explore the efficacy and safety of Pyrotinib, Trastuzumab, and Taxanes in treating Trastuzumab-treated HER2+ Advanced Breast Cancer (ABC).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old, female;
2. Pathological examination confirmed HER-2 positive invasive breast cancer; (HER2 positivity is defined as an immunohistochemical (IHC) score of 3+ or in-situ hybridization (ISH) result for HER2 gene amplification in >10% of immunoreactive cells.

   HER2 positivity needs to be verified by the pathology department of the research center involved in this study)
3. Imaging confirmed recurrent/metastatic breast cancer;
4. Patients who relapsed and metastasized three months after discontinuation of Trastuzumab treatment;
5. Have at least one measurable lesion (according to RECIST 1.1 criteria);
6. ECOG score of 0-2;
7. Expected life span ≥3 months;
8. Normal major organ function;
9. The researcher believes that the participant may benefit;
10. Volunteer to participate in this study, sign informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for participation:

1. Have any confirmed history of drug allergies, or severe allergic reactions to any component of the investigational drug (NCI-CTCAE 5.0 grade > 3);
2. Patients in advanced stages who have undergone systemic treatment;
3. A history of serious heart diseases such as congestive heart failure, unstable angina, arrhythmia or myocardial infarction;
4. Suffer from serious pulmonary diseases, such as interstitial lung disease or pneumonia, pulmonary fibrosis, acute pulmonary diseases, etc.;
5. Currently suffering from severe liver-related diseases, such as acute hepatitis, explosive hepatitis, coagulation factor synthesis disorder, etc.; Those who are positive for HBV surface antigen or HBV core antibody must have a peripheral blood Hepatitis B virus DNA titer test < 1×10 ^3 IU/ml in order to participate;
6. Comorbidity or condition that may interfere with their participation in the study, or any serious medical impediment that might affect participant's safety (such as, active or uncontrolled infection, active liver/gallbladder disease requiring antiviral treatment);
7. Other invasive tumors (including second primary breast cancer) that may affect the evaluation of results and adherence to the protocol;
8. Having undergone major surgical procedure or are yet to recover from major internal diseases within the 4 weeks prior to the study;
9. Any circumstance that the researcher considers the participant unfit to participate in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 24months
  the period of time from the start of treatment for cancer patients to the observation of disease progression, or death due to any reason

SECONDARY OUTCOMES:
CNS-PFS | 24months
  the period of time from the start of treatment for cancer patients to the observation of intracranial progression , or death due to any reason
ORR | 24months
  the proportion of patients who have a partial or complete response to therapy
DCR | 24months
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents
OS | 24months
  the period of time from the start of treatment for cancer patients to the observation of death due to any reason
Overall Number of Participants Who Experienced at Least One Adverse Event, Including Serious and Non-Serious Adverse Events | 24months
  Adverse event (AE) severity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0); if the AE was not specifically listed, the following grades of severity were used: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening or disabling; and Grade 5 = death. Severe and serious are not synonymous. Severity refers to the intensity of an AE, whereas a serious AE must meet criteria set out in the protocol; both were independently assessed for each AE. Only the most severe intensity was counted for multiple occurrences of the same AE in one participant.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No